CLINICAL TRIAL: NCT06916156
Title: A Phase 1, Open-Label, Single Center Study to Determine the Penetration of ANT3310 and Meropenem Into the Lung After Repeated Intravenous Administrations of MEM-ANT3310 in Healthy Adult Participants
Brief Title: Evaluation of the Concentration of ANT3310 and Meropenem in the Lung in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antabio (Industry)
Collaborators: Clinartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ANT3310-1003
Record Dates: First submitted 2025-04-02; First posted 2025-04-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pharmacokinetics Study on Healthy Volunteers Adults
Keywords: healthy volunteers; Bronchoalveolar lavage (BAL) study
MeSH Terms: interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ANT3310 and Meropenem (MEM) (Experimental): Each participant will receive a total of 3 doses of MEM-ANT3310, infused intravenously over 3 hours every 8 hours (i.e., 0 hour, 8 hours, and 16 hours relative to start of the first infusion).
  Interventions: Drug: ANT3310; Drug: Meropenem

INTERVENTIONS:
Drug: ANT3310 — ANT3310 will be administered in combination with Meropenem. Participants will receive 3 intravenous infusions of the combination MEM-ANT3310 every 8 hours. Infusions will be delivered through an infusion line over 3 hours at a constant rate.
Drug: Meropenem — Meropenem will be administered in combination with ANT3310. Participants will receive 3 intravenous infusions of the combination MEM-ANT3310 every 8 hours. Infusions will be delivered through an infusion line over 3 hours at a constant rate.

SUMMARY:
This is an open-label, non-randomized, single-center, repeated i.v. doses, Phase 1 trial to evaluate the pharmacokinetics, safety, and tolerability of a combination of MEM-ANT3310 in healthy adult female and male participants who will undergo a single bronchoalveolar lavage (BAL) via a standardized fiberoptic bronchoscopy to evaluate and compare the pharmacokinetics characteristics of ANT3310 and meropenem (MEM) in plasma and epithelial lining luid (ELF).

DETAILED DESCRIPTION:
There will be 25 participants enrolled in the study. Each participant will receive a total of 3 doses of MEM-ANT3310, infused intravenously over 3 hours every 8 hours. Each participant will undergo a single bronchoscopy at the assigned BAL sampling time. Blood samples will be collected. Participants will be monitored for adverse events from study center admittance through the EoS visit.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent in compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Participants must be 18 to 55 years of age, both inclusive, at the time of signing the informed consent.
* Body mass index (BMI) within the range 18.0-32.0 kg/m2 (both inclusive) and body weight > 50.0 kg (110 Ibs) at Screening.
* Contraceptive use by women or men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Healthy participants as defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, 12-lead ECG, vital signs, physical examination, spirometry at Screening (FEV1 > 80% of predicted), and clinical laboratory tests at Screening and Day -1.
* Healthy participants with vital signs at Screening and Day -1 within the normal ranges: tympanic body temperature: ≥ 35.5°C and ≤ 37.5°C; resting pulse rate ≥ 50 beats per minute (bpm) and ≤ 100 bpm; systolic blood pressure (SBP) ≥ 90 and ≤ 139 mmHg, diastolic blood pressure (DBP) ≥ 50 and ≤ 89 mmHg, taken in supine position after resting at least 5 minutes. On Day -1, blood pressure and pulse rate need to be within the normal ranges or not clinically significant range, as per investigator's judgement.
* Individualized estimated glomerular filtration rate (eGFR): [(CKD-EPI ÷ 1.73) × BSA] ≥ 90 mL/min and < 160 mL/min for males or < 150 mL/min for females at Screening.
* Sufficient venous access for i.v. infusion and PK samplings.

Exclusion Criteria:

* History of any clinically relevant gastrointestinal, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardiovascular, endocrine, hematologic, neuromuscular or allergic disease(s), metabolic disorder, cancer (may have had basal or squamous cell carcinoma of skin or cervix so long as surgically removed or deemed cured by cryotherapy, laser therapy, conization, etc, with stability for the past two years).
* History or presence of chronic pulmonary disease.
* Medical disorder, condition, or history of such that would - in the opinion of the Investigator - compromise the participant's ability to participate in this study.
* Presence of any acute illness, including febrile illness with temperature > 37.8°C (> 100.0°F), within 7 days of Baseline (Day -1 to Day 1).
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies requiring intranasal or systemic corticosteroids during any time of the year or history of any anaphylactic reaction.
* Known hypersensitivity to meropenem and or ANT3310 or any of the excipients of the infusion solution.
* Known history of clinically significant hypersensitivity or urticaria, or severe allergic reaction to β-lactam antibiotics (i.e., penicillin, cephalosporin, carbapenem, or monobactam).
* History of significant bleeding within the past 3 months.
* History of COVID-19 within three (3) months prior to Screening.
* History of epilepsy (or known seizure disorder), brain lesions or other significant neurological disorders.
* History of Gilbert syndrome.
* History of any severe antibiotic-associated superinfections, such as Clostridium difficile colitis and/or frequent fungal vaginal infections.
* Contraindications to bronchoalveolar lavage or suspected intolerability to medications necessary for bronchoscopy, hypoxemia, reactive airway disease or asthma, unstable angina or acute myocardial infarction in the last 6 months, heart failure, and severe hemostatic alterations. Anatomical or anticipated technical difficulties that would prevent bronchoscopy or BAL procedure. Allergies to lidocaine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentrations (Cmax) of ANT3310 and Meropenem after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma
Area under the concentration-time curve from 0 to 8 hours post-dose (AUC0-8h) of ANT3310 and Meropenem after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma
Percent penetration of ANT3310 and Meropenem in epithelial lining fluid (ELF) after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  ratio (%) of AUC0-8h of ELF-to-plasma for ANT3310 and Meropenem
Time from dosing to maximum observed plasma concentration (tmax) of ANT3310 and Meropenem after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) of ANT3310 and Meropenem after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma
Apparent terminal elimination half-life (t1/2λz) of ANT3310 and Meropenem in plasma after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma
Terminal phase elimination rate constant (λz) of ANT3310 and Meropenem after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma
Apparent total body clearance at steady-state (CLss) of ANT3310 and Meropenem after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma
Apparent volume of distribution at steady-state (Vss) of ANT3310 and Meropenem after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma
Apparent elimination half-life (t1/2,ELF) of ANT3310 and Meropenem in ELF after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From pre-dose to 8 hours post-last-dose
  Pharmacokinetic parameter of ANT3310 and Meropenem in ELF

SECONDARY OUTCOMES:
Number and severity of treatment-emergent adverse event (TEAE) to evaluate the safety and tolerability of ANT3310 and meropenem after repeated i.v. infusions of a combination of ANT3310 and Meropenem | From Day 1 to Day 11
  Percentage of participants experiencing ≥ one TEAE by seriousness, intensity, and relatedness from baseline through end of study visit
Number of participants who discontinue due to a TEAE. | From Day 1 to Day 11
  Percentage of participants who discontinue due to a TEAE.
Number of participants with clinically significant abnormal values for safety laboratory tests at least once post-dose | From Day 1 to Day 11
  Percentage of participants with clinically significant abnormal values for safety laboratory tests at least once post-dose
Number of participants with clinically significant abnormal values for vital signs (blood pressure, pulse rate, and body temperature) measurement at least once post-dose | From Day 1 to Day 11
  Percentage of participants with clinically significant abnormal values for vital signs (blood pressure, pulse rate, and body temperature) measurement at least once post-dose
Number of participants with clinically significant abnormal values for safety electrocardiogram (ECG) parameters at least once post-dose | From Day 1 to Day 11
  Percentage of participants with clinically significant abnormal values for safety electrocardiogram (ECG) parameters at least once post-dose
Number of infusion site reactions to assess local venous tolerability | From Day 1 to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: J. Burr Ross, MD, Principal Investigator — Pulmonary Associates, PA
Locations (1):
- Pulmonary Associates, PA, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No